CLINICAL TRIAL: NCT06946641
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effects of Single and Multiple Ascending Doses of QLS12010 Capsules in Healthy Adult Participants and Participants With Atopic Dermatitis
Brief Title: A Phase I Study of QLS12010 Capsules: Safety, Tolerability, PK, PD, and Food Effects in Healthy Adults and Moderate to Severe Atopic Dermatitis Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Qilu Pharmaceutical Research and Development Center LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLS12010-101
Record Dates: First submitted 2025-03-30; First posted 2025-04-27 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis; Hidradenitis Suppurativa (HS); Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Dermatitis, Atopic; Hidradenitis Suppurativa; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Single ascending dose cohorts in healthy participants (Experimental): Healthy volunteer subject cohorts randomized 6:2 receiving a single dose of QLS12010 or placebo. The starting dose will be 25 mg of QLS12010 or placebo.
  Interventions: Drug: QLS12010; Drug: Placebo
- Multiple ascending dose cohorts in healthy subjects (Experimental): Healthy volunteer subject cohorts randomized 8:2 to receive QLS12010 or placebo QD for 14 continuous days. The starting dose of QLS12010 or placebo is based on upcoming data from SAD part.
  Interventions: Drug: QLS12010; Drug: Placebo
- Food Effect Cohort in healthy subjects (Experimental): Part C is a two-cycle, crossover study under fasting and fed (high-fat meal) conditions. In Cycle 1, 12 healthy adult participants will be randomly divided into two groups on D-1, with 6 participants in each group receiving a single oral dose of QLS12010 Capsules under fasting or fed conditions, respectively. After completing washout, they will receive crossover administration for the Cycle 2 study.
  Interventions: Drug: QLS12010
- Early Efficacy in patients with AD (Experimental): Part D of the study plans to enroll 12 adults with moderate to severe atopic dermatitis (AD). Eligible subjects (after screening) will be sequentially assigned to two dose groups (Dose 1 and Dose 2) in the order of their enrollment. Enrollment of Dose 2 may commence only after Dose 1 has completed enrollment of 6 subjects.
  Interventions: Drug: QLS12010

INTERVENTIONS:
Drug: QLS12010 — QLS12010 oral capsule(s)
Drug: Placebo — Matching placebo oral capsule(s)
  Arms: Multiple ascending dose cohorts in healthy subjects; Single ascending dose cohorts in healthy participants

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, PK, and PD of single and multiple ascending doses of QLS12010 Capsules and the effect of food on their PK profiles in healthy adult participants and participants with atopic dermatitis. This study consists of four parts: Part A is a single ascending dose (SAD) study, once sufficient safety and PK data are obtained from the SAD cohorts, the SMC will determine the dosage of initial cohort in Part B, which consists of three multiple ascending doses (MAD) cohorts of QLS12010 Capsules. Part C is a randomized, open-label, two-cycle, crossover food effect study under fasting and fed (high-fat meal) conditions. Part D is to evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD) characteristics, and preliminary efficacy of QLS12010 Capsules following multiple oral administrations in adult participants with atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria for Parts A-C:

* Males and females aged 18-45 (inclusive),
* Weight: ≥ 50 kg for males and ≥ 45 kg for females, body mass index (BMI): 18.0-30.0 kg/m2 (inclusive),

Inclusion Criteria for Part D:

* Female or male participants between the ages of 18 to 75 years of age.
* Chronic AD diagnosed by the criteria of Hannifin and Rajka that has been present for at least 6 Months before the Screening Visit.
* At screening and baseline: EASI score ≥ 16, vIGA-AD™ score ≥ 3, and BSA affected by AD ≥ 10%;
* The weekly mean score of PP NRS ≥ 4 prior to the first administration (with assessment results for at least 4 days during the week before the first administration [D-7 to D-1]);
* As judged by the investigator, within 6 months prior to screening, the patient had an inadequate response to topical medication therapy.

General Exclusion Criteria:

* Participants with diseases that should be excluded as judged by the investigator at screening, including but not limited to the nervous system, psychiatric system, cardiovascular system, blood and lymphatic system, immune system, respiratory system, digestive system, urinary system, metabolic and skeletal system disorders,
* The 12-lead ECG at screening shows QTcF (QT corrected using Fridericia's formula) > 450 ms. If QTcF is > 450 ms, the 12-lead ECG should be repeated 2 more times (at least 3 min apart), and the mean of the 3 measurements will be used to determine whether the participant meets the inclusion criteria,
* Participants who smoke more than 5 cigarettes per day on average within 6 months before screening or are currently using e-cigarettes,
* Participants who consume more than 14 units of alcohol per week (1 unit = 360 mL of beer, 45 mL of 40% spirits, or 150 mL of wine) within 6 months before screening or have a positive breath alcohol test at screening,
* Participants who have donated more than 400 mL of blood within 3 months or more than 200 mL of blood within 4 weeks before screening, or plan to donate blood during the study,
* Participants who have received any strong inhibitor or inducer of CYP3A4 within 4 weeks before screening,
* Participants who have received any prescription drugs, OTC drugs, traditional medicines, and dietary supplements within 2 weeks before the first dose or 5 half-lives (whichever is longer).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent Adverse Events as assessed by CTCAE v5.0 | up to approximately 1 month

SECONDARY OUTCOMES:
Area under the curve plasma concentration from time zero to last measurable concentration [AUC(0-last)] | up to approximately 1 month
Area under the curve plasma concentration from time zero to infinity [AUC(0-∞)] | up to approximately 14 days
Maximum observed plasma concentration (Cmax) | up to approximately 1 month
Time to maximum observed plasma concentration (Tmax) | up to approximately 1 month
Terminal elimination half-life (t1/2) | up to approximately 1 month
Apparent clearance (CL/F) | up to approximately 1 month
Apparent volume of distribution (Vz/F) | up to approximately 1 month
Mean residence time (MRT) | up to approximately 1 month
Changes and percentage changes from baseline in Eczema Area and Severity Index (EASI) scores | at Weeks 1, 2, 3, 4, 5, and 6
  The minimum EASI score is 0, and the maximum EASI score is 72. A score of 0 indicates clear or no eczema; a greater score indicates more severe disease.
Changes and percentage changes from baseline in Investigator's Global Assessment (IGA) scale | at Weeks 1, 2, 3, 4, 5, and 6
  The IGA5-point scale ranges from 0 (clear) to 4 (severe AD). A decrease in score indicates an improvement in signs and symptoms.
Changes and percentage changes from baseline in weekly mean scores of Peak Pruritus Numerical Rating Scale (PP NRS) | at Weeks 1, 2, 3, 4, 5, and 6
  The PP NRS is a single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 h based on the following question: 'On a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable".
Changes and percentage changes from baseline of body surface area (BSA) affected by lesions | at Weeks 1, 2, 3, 4, 5, and 6
  BSA assessment estimates the area of skin lesions in each part of the body, with one palm unit of the patient taken as 1% of the body surface area.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China